CLINICAL TRIAL: NCT00792090
Title: Use of Fermented Milk in Prevention of Cow's Milk Allergy in New Born and Infant
Brief Title: Prevention of Cow's Milk Allergy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bledina (Industry)
Collaborators: Optimed Medizinische Instrumente GmbH (Industry)
Responsible Party: Valérie BRENAS, Bledina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BL006
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Milk Hypersensitivity
Keywords: allergy; cow's milk; sensibilisation; fermented milk; infant formula
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fermented milk
  Interventions: Other: Fermented milk
- 2 (Active Comparator): Standard milk
  Interventions: Other: Standard milk

INTERVENTIONS:
Other: Fermented milk — Formula used for non breastfed children or in complement of breastfeeding
  Arms: 1
Other: Standard milk — Formula used for non breastfed children or in complement of breastfeeding
  Arms: 2

SUMMARY:
Impact of fermented milk in prevention of cow's milk allergy in new born and infants

ELIGIBILITY:
Inclusion Criteria:

* mother before the 5th month of pregnancy
* mother agreeing to stop consumption of yogurts and fermented milks during the 3rd quarter of pregnancy
* mother agreeing to receive a calcium supplementation during the 3rd quarter of pregnancy
* atopic mother or father and at least another atopic member (sister or brother)
* parents having given written informed consent
* adhesion to eviction regimen for mother and child
* parents agreeing with a regular follow-up (3 visits and monthly phone call with the dietician)

Exclusion Criteria:

* mother in an exclusion period from another study
* parents refusing to sign the informed consent
* infant in a situation which could interfere with an optimal participation to the study, or which could represent a risk for the infant, according to the investigator
* known or suspected immunodeficiency in the family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2003-11; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Sensibilisation and cow's milk allergy | 4, 12 and 24 months

SECONDARY OUTCOMES:
Sensitization or allergy to other allergens | 4, 12 and 24 months
Atopic diseases (atopic dermatitis, asthma) | 4, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dupont, PhD, Principal Investigator — Hôpital Saint Vincent de Paul; Denise-Anne Moneret-Vautrin, PhD, Principal Investigator — Hôpital central
Locations (2):
- France (2):
  - Hôpital central, Nancy
  - Hôpital Saint Vincent de Paul, Paris